CLINICAL TRIAL: NCT01186198
Title: A Clinical Evaluation of the MINI TREK RX 1.20 mm Coronary Dilatation Catheter in Stenotic Lesions
Acronym: CROSS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-802
Record Dates: First submitted 2010-08-09; First posted 2010-08-23 (Estimated); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Heart Disease; Coronary Artery Stenosis; Chronic Coronary Total Occlusion; Coronary Bypass Graft Stenosis
Keywords: Coronary Dilatation Catheter; Balloon Dilatation Catheter; Angioplasty; Myocardial Ischemia; Coronary Stenosis; Percutaneous Coronary Intervention (PCI); Percutaneous Transluminal Coronary Angioplasty (PTCA); Chronic Total Occlusion (CTO)
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- MINI TREK RX 1.20 mm Coronary Dilatation Catheter: Patients requiring initial balloon dilatation of the stenotic portion of a coronary artery or bypass graft stenosis will be included.
  Interventions: Device: MINI TREK RX 1.20 mm Coronary Dilatation Catheter

INTERVENTIONS:
Device: MINI TREK RX 1.20 mm Coronary Dilatation Catheter — Enlarging coronary luminal diameter during percutaneous coronary intervention (PCI) procedures in subjects with ischemic heart disease due to stenotic lesions

SUMMARY:
This is a prospective, single-arm, open-label, multi-center, observational study to assess the acute safety and efficacy of MINI TREK RX 1.20 mm for enlarging coronary luminal diameter during percutaneous coronary intervention (PCI) procedures in subjects with ischemic heart disease due to stenotic lesions.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedure.
3. Subject must have stenotic lesion(s) in native coronary arteries or bypass grafts that are suitable for percutaneous coronary intervention.
4. Subject must have single or multiple vessel coronary artery disease with clinical evidence of myocardial ischemia (e.g., stable or unstable angina or silent ischemia documented by a positive functional study).
5. Subject must be an acceptable candidate for CABG.
6. Subject must agree to undergo all protocol-required follow-up procedures.
7. Subject must agree not to participate in any other clinical study during hospitalization for the index procedure.

Angiographic Inclusion Criteria

All angiographic inclusion criteria are based on visual estimation.

1. De novo or restenotic lesions in native coronary arteries or bypass grafts.
2. A maximum of two lesions, including at least one target lesion, in up to two major epicardial distribution trees. Tandem lesions, defined as multiple, focal lesions that can be covered by one stent, will be considered as a single lesion.
3. If one target lesion and one non-target lesion are to be treated, the target and non-target lesions must be located in different major epicardial distribution trees.
4. The target lesion must have a diameter stenosis of ≥ 70% by visual estimation or online quantitative coronary angiography (QCA), which may include chronic total occlusion (CTO).
5. Lesions may be located in highly tortuous vessels.

Exclusion Criteria:

General Exclusion Criteria

1. Subject has had a known diagnosis of an acute myocardial infarction (AMI) within 72 hours preceding the intended index procedure.
2. The subject is currently experiencing clinical symptoms consistent with a new onset of AMI, such as prolonged chest pain with ischemic ECG changes unresponsive to nitrates.
3. Subject has hemodynamic instability or any hemodynamically unstable cardiac arrhythmias.
4. Subject has a known left ventricular ejection fraction (LVEF) < 30% at the most recent evaluation (LVEF may be obtained at the time of the index procedure if the value is unknown and if necessary).
5. Subject is receiving chronic anticoagulation therapy (e.g., heparin, coumadin).
6. Subject will require Low Molecular Weight Heparin (LMWH) within 8 hours before or at any time after the index procedure.
7. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, anti-platelet medications, or sensitivity to contrast media, which cannot be adequately pre-medicated.
8. Subject has a platelet count < 100,000 cells/mm^3 or > 700,000 cells/mm^3.
9. Subject has a serum creatinine level > 2.0 mg/dl within seven days prior to index procedure.
10. Subject has had a cerebrovascular accident/stroke or transient ischemic neurological attack (TIA) within the past six months.
11. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
12. Subject has had active peptic ulcer or a significant gastrointestinal or urinary bleed within the past six months.
13. Elective surgery is planned during hospitalization for the index procedure that will require discontinuing dual anti-platelet therapy.
14. Subject has other medical illness (e.g., cancer) that may confound the data interpretation or is associated with a limited life expectancy.
15. Subject is currently participating in an investigational study when such participation could confound the treatment or outcomes of this study.
16. Subject is pregnant or nursing. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Angiographic Exclusion Criteria

All angiographic exclusion criteria are based on visual estimation.

1. More than two lesions require treatment. Tandem lesions, defined as multiple, focal lesions that can be covered by one stent, will be considered as a single lesion.
2. Target lesion is located in an unprotected left main artery.
3. Coronary artery spasm in the absence of significant stenosis.
4. Target vessel contains thrombus as indicated in the initial angiographic images.
5. During the index procedure, any lesion requires additional treatment with any adjunctive or ablative device (i.e., rotational or directional atherectomy, cutting balloon, laser, thrombectomy, etc.).
6. Target lesion involving a bifurcation with a side branch ≥ 2.5 mm in diameter, with an ostial lesion > 40% stenosed, or with a side branch requiring protection guide wire or pre-dilatation.
7. Additional clinically significant lesion(s) in any coronary arteries or bypass grafts for which PCI may be required during hospitalization for the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled at 4 sites in the United States (US). At each site, at least two different qualified physicians will perform the index procedures. Approximately 30% of the enrolled subjects will be females.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2010-12-30 (Actual); Study Completion 2010-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (4):
- United States (4):
  - Scripps Green Hospital, La Jolla, California
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Northern Michigan Hospital, Petoskey, Michigan
  - The Christ Hospital, Cincinnati, Ohio

REFERENCES:
- [Derived] Kandzari DE, Teirstein PS, Kereiakes DJ, Cannon LA, Hearne SE, Kuo HC, Ying SW, Cheong WF, Popma JJ. Procedural effectiveness of a novel 1.20 mm diameter angioplasty catheter: clinical and angiographic outcomes. J Interv Cardiol. 2013 Apr;26(2):131-6. doi: 10.1111/j.1540-8183.2013.12021.x. Epub 2013 Jan 31. PMID 23369084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 subjects were enrolled at 4 clinical sites in the US between August 12, 2010 and December 30, 2010. All subjects were followed in-hospital up to discharge.
Period: Overall Study
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 71 patients were enrolled; however, subjects can be counted in more than one race category therefore the total in the table by race is greater than 71 patients.
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.75 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  American Indian or Alaskan Native | 0
  Asian | 2
  Black or African Heritage | 2
  Native Hawaiian or Pacific Islanders | 0
  White | 68
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71
Prior coronary intervention [Count of Participants; unit: Participants] | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Procedure Success
Description: Procedure success was defined as meeting all the following after single or multiple attempts:
  1. Successful delivery of the MINI TREK RX 1.20 mm balloon to and across the target lesion,
  2. Successful inflation and deflation with the MINI TREK RX 1.20 mm balloon,
  3. No vessel perforation, no flow-limiting vessel dissection, no reduction in TIMI flow from baseline, and no clinically significant arrhythmias requiring medical treatment or device intervention following dilatation with the MINI TREK RX 1.20 mm balloon, and
  4. Achieve a final TIMI flow grade of 3 at the conclusion of the PCI procedure for the lesion.
Time Frame: On Day 0 (From the start to end of the interventional procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 67
percentage of participants | 98.5 [91.96 to 99.96]

2. Secondary Outcome: Rate of Device Success
Description: Device Success was defined as meeting all the following after single or multiple attempts:
  1. Successful delivery of the MINI TREK RX 1.20 mm balloon to and across the target lesion, defined as achieving a final residual percent diameter stenosis of < 50%,
  2. Successful dilatation with the MINI TREK RX 1.20 mm balloon as defined by improvement in Minimal Lumen Diameter (MLD) based on core lab analysis, and
  3. No vessel perforation, no flow-limiting vessel dissection, no reduction in TIMI flow from baseline, and no clinically significant arrhythmias that required medical treatment or device intervention following dilatation with the MINI TREK RX 1.20 mm balloon.
Time Frame: On Day 0 (From the start to end of the interventional procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: Percentage of target lesions
Units Other Than Participants: Target lesions
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 71
Number analyzed (Target lesions) | 78
Percentage of target lesions | 96.2 [89.17 to 99.20]

3. Secondary Outcome: Rate of Lesion Success
Description: Lesion Success was defined as meeting all the following after single or multiple attempts:
  1. Successful dilatation with any device(s), defined as achieving a final residual percent diameter stenosis of < 50%,
  2. No vessel perforation, no flow-limiting vessel dissection, no reduction in TIMI flow from baseline, and no clinically significant arrhythmias requiring medical treatment or device intervention following dilatation with any device(s), and
  3. Achievement of a final TIMI flow grade of 3 at the conclusion of the PCI procedure for the lesion.
Time Frame: On Day 0 (From the start to end of the interventional procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number (95% Confidence Interval); unit: Percentage of target lesions
Units Other Than Participants: Target lesions
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 71
Number analyzed (Target lesions) | 83
Percentage of target lesions | 97.6 [91.57 to 99.71]

4. Secondary Outcome: Rate of Individual Procedural Parameters
Description: The following parameters were assessed by either an angiographic core laboratory or the investigator at the site
  * Vessel perforation
  * Flow-limiting vessel dissection
  * Development of thrombus in the target vessel
  * Balloon rupture
  * Clinically significant arrhythmias requiring medical treatment or device intervention
Time Frame: On Day 0 (From the start to end of the interventional procedure)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 71
Number analyzed (Target lesions) | 83
percentage of participants
  Vessel Perforation | 0.0
  Flow-Limiting Vessel Dissection | 0.0
  Development of Thrombus in the Target Vessel | 0.0
  Balloon Rupture | 0.0
  Clinically Significant Arrhythmias Requiring Medical Treatment or Device Intervention | 0.0

5. Secondary Outcome: Rate of Major Adverse Cardiac Event (MACE)
Description: In-hospital MACE was defined as the composite of all deaths, myocardial infarction (MI), and clinically indicated target lesion revascularization (CI-TLR) by coronary artery bypass graft surgery (CABG) or PCI during the hospitalization for the index procedure
Time Frame: In-Hospital (1 - 3 Days)
Population: The number of participants analyzed includes subjects who were available at that timeof analysis
Measure: Count of Participants; unit: Participants
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 71
Participants | 6

6. Secondary Outcome: Rate of Target Lesion Failure (TLF)
Description: In-hospital TLF was defined as the composite of cardiac death, target vessel myocardial infarction (TV-MI), and CI-TLR by CABG or PCI during the hospitalization for the index procedure
Time Frame: In-Hospital (1 - 3 Days)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 71
Participants | 6

7. Secondary Outcome: Rate of Stent Thrombosis
Description: Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation.
  Angiographic confirmation involves presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent and presence of at least 1 of the following criteria within 48-hours:
  Acute onset of ischemic symptoms at rest; New ischemic ECG changes that suggest acute ischemia; Typical rise and fall in cardiac biomarkers; Non-occlusive; Occlusive thrombus
  Evidence of recent thrombus within the stent determined at autopsy or via examination of tissue retrieved following thrombectomy is a pathological confirmation.
  Probable stent thrombosis is considered to have occur after intracoronary stenting in case of any unexplained death within the first 30 days or any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: In-Hospital (1 - 3 Days)
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
Number analyzed (Participants) | 64
percentage of participants
  Acute Stent Thrombosis | 0
  Subacute Stent Thrombosis | 0
  Acute/Subacute Stent Thrombosis | 0

ADVERSE EVENTS:
Time Frame: In-hospital Assessment Only
Arm/Group | MINI TREK RX 1.20 mm Coronary Dilatation Catheter
All-Cause Mortality (participants affected / at risk) | 0/71
Serious Adverse Events (participants affected / at risk) | 6/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MINI TREK RX 1.20 mm Coronary Dilatation Catheter (N=71)
Periprocedural Non-Q-wave Myocardial Infarction (NQMI) (Cardiac disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days